CLINICAL TRIAL: NCT07225218
Title: Targeted Upstream Prevention (T-UP): Engaging Vulnerable Students in Diabetes Prevention
Brief Title: New T-UP: Engaging Vulnerable Students in Diabetes Prevention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Principal Investigator, Lauren Wisk, PhD, Assistant Professor, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: IRB#25-1605
Record Dates: First submitted 2025-11-04; First posted 2025-11-06 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-07

CONDITIONS: Prediabetes; Type 2 Diabetes
MeSH Terms: conditions — Prediabetic State; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diabetes Prevention Program (DPP) group (Experimental): The DPP group will receive a tailored Diabetes Prevention Program. The DPP group will complete intervention lessons online and asynchronously. Each lesson typically takes on average 15 minutes to complete.
  Interventions: Behavioral: Tailored DPP Intervention
- Control group (No Intervention): The control group will receive access to a study habits intervention (fall), alcohol use intervention (winter), and financial literacy intervention (spring). The control group will receive each intervention materials via e-mail for participants to review on their own time. The interventions for the control group will be remote. A research assistant will meet with control participants via Zoom to explain the intervention materials. The Zoom session will take approximately 1 hour.

INTERVENTIONS:
Behavioral: Tailored DPP Intervention — The DPP intervention will be online and asynchronously. Participants will be asked to complete the intervention lessons on their own time. Each lesson typically takes on average 15 minutes to complete.
  Arms: Diabetes Prevention Program (DPP) group

SUMMARY:
The goal of this study is to enhance reach and uptake of diabetes prevention among young adults, with a focus on recruiting underserved and high-need students who face additional challenges, including food and financial insecurity.

The specific aims are:

Aim 1 - Evaluate the efficacy of an AYA-tailored version of the UC DPP for mitigating type 2 diabetes risk (i.e., weight change) in a pre/post pilot trial. The investigators hypothesize that the AYA-tailored intervention will be effective at producing 5% weight loss from baseline to program completion (at 9-months).

Aim 2 - Assess the feasibility and acceptability of an AYA-tailored version of the UC DPP program. The investigators hypothesize that it will be feasible to recruit the desired number of participants given proposed innovative outreach strategies, and that the AYA-tailored intervention will be deemed acceptable to participants both qualitatively and in regards to their retention in the program at rates similar to the larger UC DPP.

The investigators will recruit 80 UCLA undergraduate students. Participants will be asked to complete a brief screening online form to assess eligibility and to collect contact information. The PI and/or Research Assistants (RAs) will reach out to eligible participants to obtain informed consent and enroll them in the pilot trial. The investigators will randomize participants to the tailored DPP cohort vs control cohort. Control participants will be offered the opportunity to participate in the tailored DPP in the following academic year. The tailored DPP intervention will be online and asynchronously. Participants will be asked to complete the intervention lessons on their own time. Each lesson typically takes on average 15 minutes to complete.

Control group will receive each intervention materials via e-mail for participants to review on their own time and will receive acceptability surveys. The interventions for the control group will be remote. A research assistant will meet with control participants via Zoom to explain the intervention materials. Control group will receive access to a study habits intervention, alcohol use intervention, and financial literacy intervention.

At the end of each quarter (Fall, Winter, and Spring), both control and intervention participants will receive an email with a unique link to a brief REDCap survey to ascertain acceptability of sessions/lessons.

Furthermore, participants will complete baseline and 9-month follow-up assessments. Participants will complete a 30 minute questionnaire and height/weight measurements will be collected by a RA. Participants will be asked to self-report weight and physical activity at the end of the fall and winter quarter; data will be collected via brief REDCap survey.

DETAILED DESCRIPTION:
Aim 1 - Design: Pre/post pilot trial of 80 participants (<1% of total number of eligible UCLA undergraduates). The investigators will randomize participants to the tailored DPP vs control based on a stratified, block (n=2) schema based on age [≤19/≥20] and sex [M/F]. All control participants will be offered the opportunity to participate in the tailored DPP in the following academic year (in the interest of equipoise).

Aim 1 - Participant Recruitment: All participants will be asked to complete a brief screening online form to assess eligibility and to collect contact information. This form will further allow us to prioritize recruitment efforts of those with identified food, financial, or stress-related vulnerability. After confirming eligibility, a trained research assistant (RA) will reach out to eligible participants to obtain informed consent and enroll them in the pilot trial.

Aim 1 - Tailored DPP Intervention: Once consented and enrolled, participants will be randomized into one of two cohorts, the first group will be enrolled in the tailored DPP for the immediate academic year while the second will be enrolled in a series of unrelated interventions in year 1 and offered the opportunity to participate in the tailored DPP for the following academic year. The tailored DPP intervention will be online and asynchronously. Participants will be asked to complete the intervention lessons on their own time. Each lesson typically takes on average 15 minutes to complete.

The control group will receive access to a study habits intervention (fall), alcohol use intervention (winter), and financial literacy intervention (spring).

The control group will receive each intervention materials via e-mail for participants to review on their own time. The interventions for the control group will be remote. A research assistant will meet with control participants via Zoom to explain the intervention materials. The Zoom session will take approximately 1 hour. There will be three zoom sessions in total (one for each intervention). At the end of each quarter (Fall, Winter, and Spring), control participants will receive an email with a unique link to a brief REDCap survey to ascertain acceptability of the sessions. The acceptability survey that will be sent to participants at the end of Fall and Winter quarters will ask participants to rate satisfaction of the sessions that they completed/attended during the quarter on a 5-point Likert scale ("very dissatisfied" to "very satisfied") with respect to a) content, b) coach, c) group interaction, and d) overall, and to self-report their weight and physical activity.

Aim 1 - Data Collection: Participants will complete two study assessments (baseline and 9-month follow-up). There are two assessments per year, baseline and 9-month follow up for the first year and baseline and 9-month follow-up for the second year. These assessments will be done around October and June, respectively. Participants will complete a 30-minute questionnaire (administered as a REDCap survey) and height/weight measurements will be collected using a standardized protocol by a trained research assistant. RA will meet participants in the Wooden Center at UCLA to collect measurements. Participants will be asked to self-report weight and physical activity at the end of the fall and winter quarter; data will be collected via brief REDCap survey.

Furthermore, if participants can't attend the baseline and 9-month follow-up height/weight measurements in-person appointments. Participants will be asked to share their height/weight measurements via email. If they had a recent healthcare appointment, or if they have any doctor's visits planned, participants will be asked to submit a photo of their height and weight measurements that were taken at their doctor's visit or a printout (like an after-visit summary) with their height/weight from the doctor. If they don't have any doctor's appointments, participants will be asked to submit a photo of them taking their own height and weight measurements at home.

Aim 1 - Measures: The baseline survey assessment will collect data using validated tools on sociodemographics (e.g., age, sex, race, ethnicity, socioeconomic status), social vulnerability (food security using the USDA ERS Food Security 6-Item Short Form, financial security using the Financial Chronic Stress Scale), health-related quality of life (CDC's HRQoL tool), mental health (depressive symptoms via Patient Health Questionnaire-8; anxiety symptoms via Generalized Anxiety Disorder-7), self-perceived weight status (How do you describe your weight?), and self-reported physical activity and diet (using the International Physical Activity Questionnaire and Nutrition Screening Survey). The follow-up survey assessment (at 9 months) will collect data on health-related quality of life, mental health, self-perceived weight status, and self-reported physical activity and diet. At both time points, height and weight data will be collected by a trained research assistant.

Aim 2 - Design: Longitudinal analysis of participants of the treatment arm (N=40 in the tailored DPP cohort).

Aim 2 - Data Collection: At the end of each quarter (Fall, Winter, and Spring), participants will receive an email with a unique link to a brief REDCap survey to ascertain acceptability of the lessons. The acceptability survey that will be sent to participants at the end of Fall and Winter quarters will ask participants to rate satisfaction of the lessons that they completed during the quarter on a 5-point Likert scale ("very dissatisfied" to "very satisfied") with respect to a) content, b) coach, and c) overall, and to self-report their weight and physical activity. The investigators will implement targeted follow-up reminder schemes via text-messaging and/or e-mail, to improve participant response rates to these brief assessments.

Aim 2 - Measures: To assess feasibility the investigators will determine proportion of participants who are recruited (enrolled/those completing the initial screen) and retained (lesson completion/enrolled). Recruitment source (student health referral vs diffuse outreach/self-referral) will be compared to determine if characteristics of participants differed by recruitment source. Acceptability surveys will ask participants to rate satisfaction of the quarterly lessons on a 5- point Likert scale ("very dissatisfied" to "very satisfied") with respect to a) content, b) coach, and c) overall. Surveys will include an open-ended question to elicit participants' specific thoughts/perspectives on quarter's lessons (Fall, Winter, and Spring). Retention will be ascertained by intervention staff.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are currently enrolled (either full time or part time) as an undergraduate at UCLA and meet criteria for the T-UP Wellness Program (students who have a BMI of ≥25 (≥23 for those self- identifying as Asian) and either documented prediabetes or identified as high-risk on a CDC questionnaire).

Exclusion Criteria:

* Participants who are not currently enrolled (either full time or part time) as an undergraduate at UCLA and do not meet criteria for the T-UP Wellness Program.

Ages: 17 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-10-14 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Change in weight (pounds, lbs) between baseline and 9-month follow-up | 9 months
  A physical scale will be used to assess the percent weight (in pounds) at baseline and at 9-months follow-up; change in these two measures will be calculated and used as the primary outcome. The investigators are comparing the percentage change between participants' final weight (in pounds) measurement versus baseline weight (in pounds) measurement as a fraction of participants' baseline weight measurement (= (final - baseline) / baseline)).
Change in self-reported quality of life (Centers for Disease Control and Prevention Health-Related Quality of Life-14 item (CDC HRQOL-14)) between baseline and 9-month follow-up | 9 months
  A self-reported questionnaire will be administered at baseline and 9-month follow-up and will include questions from the three different modules of the CDC HRQOL-14. The summary "unhealthy days" index, which ranges from 0-30 unhealthy days, will be calculated. Higher scores indicate worse health/well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren E Wisk, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will add data resources on the UCLA Dataverse, a general data repository, or equivalent. The data repository will include the data codebook and information to submit a reasonable request for data access. Reasonable request will be one that meets the following criteria: submitted by a credentialed (professional/graduate degree holder or student) researcher affiliated at a college, university, medical center/system or other non-profit institution, with a proposed research question that is addressable with the available data (regardless of the perceived merit of the question), who is willing to agree to cite the original data source and ADA as a funding source for all research products using the data, and who is willing to agree to not attempt to identify any of the participants included in the dataset. Once a reasonable request has been submitted, the investigators will provide aggregate, de-identified study data to researchers.
Time Frame: The data dictionary/codebook and request instructions will be made available 6 months after the completion of data collection and cleaning.
Access Criteria: A credentialed researcher affiliated at a college, university, medical center/system or other non-profit institution, with a proposed research question that is addressable with the available data, who is willing to agree to cite the original data source and ADA as a funding source for all research products using the data, and who is willing to agree to not attempt to identify any of the participants included in the dataset.